CLINICAL TRIAL: NCT00667680
Title: Transcranial Direct Current Stimulation (tDCS) in Treatment-resistant Depression - Effect on Clinical and Neurophysiological Parameters
Brief Title: Transcranial Direct Current Stimulation (tDCS) in Treatment-resistant Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Frank Padberg, MD, PhD, Dept. of Psychiatry, Ludwig-Maximilians-University Munich
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01/2007
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Last update posted 2009-11-16 (Estimated); Status verified 2009-11

CONDITIONS: Therapy Resistant Major Depression
Keywords: tDCS, major depression
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): anodal tDCS
  Interventions: Device: Transcranial direct current stimulation (tDCS) - Eldith DC-Stimulator
- 2 (Sham Comparator): Sham tDCS
  Interventions: Device: Transcranial direct current stimulation (tDCS) - Eldith DC-Stimulator

INTERVENTIONS:
Device: Transcranial direct current stimulation (tDCS) - Eldith DC-Stimulator — real or sham tDCS for 20 minutes at 2mA intensity over the left DLPFC (F3 according to the 10-20 system)
  Other Names: Eldith DC - Stimulator (neuroConn GmbH, Ilmenau, Germany)

SUMMARY:
tDCS applies a small amount of direct electric current (DC) to the brain by means of two electrodes: the one is an active electrode, localized on the effective site, and the other is a reference electrode, localized on some "silent" part of the body. Anodal transcranial direct current stimulation (tDCS) of the left dorsolateral prefrontal cortex (DLPFC) has been associated with working memory enhancement and improvement of mood. This study will investigate the possible antidepressant effects of tDCS in patients with therapy resistant major depressive episodes.

DETAILED DESCRIPTION:
Transcranial direct current stimulation (tDCS) is a non-invasive method that shifts membrane potential towards hypo- or hyperpolarization and therefore leads to functional changes in a discrete area of the cerebral cortex.

Neurophysiological studies have shown that slow changes in cortical scalp potential reflect overall activity of cortical neuronal networks. These scalp potentials reflect shifts in membrane potentials of the cortical neurons. Over the past 7 years tDCS has evolved as an important tool to non-invasively manipulate specific neural circuits of the human brain.

The purpose of this study is an investigation of tDCS applied to 20 therapy-resistance major depressive patients. Our hypothesis is that tDCS may exert an antidepressant effect and/or enhances the medication effect. tDCS will be examined in the framework of a placebo-controlled clinical pilot-study investigating effectiveness, safety and influence on EEG parameters. Patients will receive anodal DC stimulation or sham stimulation (extra designed placebo-stimulator) in a double-blind design over 10 days for each condition. Outcomes will be evaluated using several clinical, psychiatric and neuropsychological rating scales.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* At least moderate major depressive episode (DSM IV criteria).
* Stable total pre-treatment Hamilton Rating Scale for Depression score ≥18
* Therapy-resistance during current depressive episode (according to ATHF).
* The patient must be in the condition to understand the patient-information, as well as the necessary examinations. He/she must be able to give a written consent.
* Stable antidepressant medication, that is retained during the study- duration, from at least three weeks before the begin of the study.

Exclusion Criteria:

* Existence of a care/legal incapacity
* Existing pregnancy
* Severe psychiatric illness (with exception of affective disorder)
* Acute suicidality
* Drug-, medication- or alcohol dependence
* Dementia according to DSM IV / ICD 10-criterions
* Severe TBI in the anamnesis
* Indications of structural damage of the basal ganglia or the brain stem
* Severe neurological disorders (e.g. M. Parkinson, epilepsy, discus-prolapse, dementia, systemic neurological illnesses, normal pressure hydrocephalus, cerebrovascular diseases, elevated intracranial pressure, in the last 6 months, polyneuropathies).
* Severe other medical conditions, like manifest arterial hypertonia, severe heart disease, pacemakers, respiratory failure, malignant illnesses all type, also in the history, active infectious diseases, skeletal disorders (like M. Paget, osteoporosis with spontaneous fractures, fresh fractures)
* Other circumstances, that speaks against a participation of the patient pinion of MD at this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-03; Primary Completion 2008-09 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Hamilton Psychiatric Rating Scale for Depression (HRSD-24) | 6

SECONDARY OUTCOMES:
Beck depression Inventory (BDI) Clinical Global Impression (CGI) Mini-Mental-Status-Test (MMST) Verbal Learning and Memory Test (VLMT) Regensburger Word Fluency Test (RWT) | 4

CONTACTS AND LOCATIONS:
Overall Officials: Frank Padberg, MD, PhD, Principal Investigator — Dept. of Psychiatry, Ludwig-Maximilians-University Munich
Locations (1):
- Department of Psychiatry and Psychotherapy, Ludwig-Maximilian University Munich, Munich, Germany

REFERENCES:
- See also: Related Info — http://psywifo.klinikum.uni-muenchen.de/forschung/tms/indexeng.html